CLINICAL TRIAL: NCT00670761
Title: Misoprostol for the Treatment of Incomplete Abortion: Comparison of Treatment Options
Brief Title: Misoprostol for the Treatment of Incomplete Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Befelatanana Maternity Centre (Unknown); Municipal Clinical Hospital No. 1 (Unknown); Kagera Regional Hospital (Other); Jose Macamo Hospital (Unknown); Tudu hospital (Unknown); National OBGYN hospital (Unknown); Cuchi General District hospital (Unknown); Hôpital de District Sanitaire Dandé (Unknown); Hôpital de District Sanitaire de Ziniaré (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2.2.1
Record Dates: First submitted 2008-04-29; First posted 2008-05-02 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Abortion, Incomplete
Keywords: misoprostol; incomplete abortion; sublingual; postabortion care; MVA
MeSH Terms: conditions — Abortion, Incomplete | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): treatment with 600mcg oral misoprostol
  Interventions: Drug: misoprostol
- 2 (Active Comparator): treatment with 400mcg sublingual misoprostol
  Interventions: Drug: misoprostol
- 3 (Active Comparator): treatment with Manual Vacuum Aspiration (MVA)
  Interventions: Procedure: MVA

INTERVENTIONS:
Drug: misoprostol — comparison of orally administered 600mcg of misoprostol to either sublingually administered 400mcg or Manual Vacuum Aspiration (MVA)
  Other Names: Cytotec
  Arms: 1; 2
Procedure: MVA — comparison of orally administered 600mcg of misoprostol to either sublingually administered 400mcg or Manual Vacuum Aspiration (MVA)
  Arms: 3

SUMMARY:
This randomized study will examine the efficacy, safety and acceptability of misoprostol for treatment of incomplete abortion.

Women diagnosed with incomplete abortion will be randomized to receive one of the following regimens:

In Tanzania and Mozambique:

1. 600 mcg of oral misoprostol in one dose, or
2. Standard surgical treatment (MVA)

In Moldova and Madagascar:

1. 600 mcg of oral misoprostol in one dose, or
2. 400 mcg of sublingual misoprostol in one dose.

In Burkina Faso and Vietnam:

1. 400 mcg of sublingual misoprostol in one dose.

We hypothesize that treatment of incomplete abortion with either 400 mcg sublingual misoprostol, 600 mcg oral misoprostol or MVA are equally effective in evacuating the uterus.

ELIGIBILITY:
Inclusion Criteria:

* If no ultrasound used:

  1. Past or present history of vaginal bleeding during pregnancy; and
  2. Open cervical os.
* If ultrasound used:

  1. Past or present history of vaginal bleeding during pregnancy; and
  2. Evidence of incomplete abortion with substantial debris in the uterus.

All women would have been advised to have surgical evacuation of the uterus if misoprostol was not available.

* Willing to provide contact information for purposes of follow-up.

  * In Tanzania: 18 years of age or over or parental permission
  * In Mozambique: 21 years of age or over or parental permission
  * In Moldova: 18 years of age or over
  * In Madagascar: 18 years of age or parental permission
  * In Vietnam: reproductive age

Exclusion Criteria:

* Contraindications to the study drug;
* Uterine size larger than 12 weeks L.M.P. at time of presentation for care.
* Signs of severe infection, defined as at least one of the following of:

  1. foul smelling discharge,
  2. fever > 39 degrees C ,
  3. pulse >110/min;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2004-07; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
complete resolution of signs/symptoms of incomplete abortion without recourse to surgery at any point for any reason | one week after initial treatment with the option of an additional week

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (6):
- Burkina Faso (2):
  - Hôpital de District Sanitaire Dandé, Bobo-Dioulasso
  - Hôpital de District Sanitaire de Ziniaré, Ouagadougou
- Befelatanana Maternity Centre, Antananarivo, Madagascar
- Municipal Clinical Hospital, Chishinau, Moldova
- Jose Macamo Hospital, Maputo, Mozambique
- Kagera Regional Hospital, Bukoba, Tanzania

REFERENCES:
- [Derived] Ngoc NT, Shochet T, Blum J, Hai PT, Dung DL, Nhan TT, Winikoff B. Results from a study using misoprostol for management of incomplete abortion in Vietnamese hospitals: implications for task shifting. BMC Pregnancy Childbirth. 2013 May 22;13:118. doi: 10.1186/1471-2393-13-118. PMID 23697561